CLINICAL TRIAL: NCT04865679
Title: Tolerability and Feasibility Pilot Clinical Study of a Large-Diameter Nerve Cap for Protecting and Preserving Terminated Nerve Ends
Acronym: REPOSE-XL℠
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP-CP-002; CDMRP-OR180222 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-04-22; First posted 2021-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Symptomatic Neuroma; Amputation; Chronic Nerve Pain
Keywords: Peripheral Nerve Injuries; Peripheral Nervous System Disease; Neuroma; Nerve Pain; Nervous System Diseases; Trauma - Nervous System; Amputation; Nerve Repair; Surgical Treatment of Pain
MeSH Terms: conditions — Peripheral Nerve Injuries; Peripheral Nervous System Diseases; Neuroma; Neuralgia; Nervous System Diseases; Trauma, Nervous System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Axoguard Nerve Cap® (Experimental): Active Comparator: Porcine derived extracellular matrix (ECM) based Nerve Termination Device
  Implantation of appropriate diameter of Axoguard Nerve Cap® (sizes 5-7 mm) at the time of surgery
  Interventions: Device: Axoguard Nerve Cap®

INTERVENTIONS:
Device: Axoguard Nerve Cap® — Entubulation of the nerve stump into the Axoguard Nerve Cap® following surgical excision of symptomatic neuroma

SUMMARY:
This pilot study evaluates the tolerability and feasibility of the Axoguard Large-Diameter Nerve Cap (sizes 5-7 mm) for protecting and preserving terminated nerve endings after limb trauma or amputation when immediate attention to the nerve injuries is not possible.

ELIGIBILITY:
Inclusion Criteria: Potential Subjects MUST:

1. Sign and date an IRB-approved written Informed Consent Form prior to initiation of any study procedures;
2. Be an adult male or female ≥ 18 and ≤ 80 years of age;
3. Present for surgery with either:

   1. Limb trauma and/or planned amputation of a limb and be candidates who are planned for a secondary nerve surgery such as Targeted Muscle Reinnervation (TMR) or Regenerative Peripheral Nerve Interface (RPNI) procedures within 6-12 months from time of amputation, or;
   2. A previous amputation and be undergoing surgery to address nerve ends;
4. Have at least one nerve end measuring greater than 4 mm and less than 7 mm in diameter after debridement and hemostasis of the proximal nerve stump;
5. Have sufficient soft tissue available to be adequately covered by the Axoguard Nerve Cap;
6. Be willing and able to comply with all aspects of the treatment and follow-up assessments and to return for all required study visits throughout the study duration.

Exclusion Criteria: Potential Subjects MUST NOT:

1. Currently undergoing or are expected to undergo treatment with chemotherapy, radiation therapy, or other known treatment that affects the growth of neural and/or vascular tissues;
2. Have signs and symptoms of chemotherapy-induced peripheral neuropathy from previous chemotherapy;
3. Be immunosuppressed or have planned immunosuppressive therapy during the duration of the study;
4. Current uncontrolled local or systemic infection as indicated by positive blood culture or other pathological indicators of infection;
5. Be contraindicated for soft tissue implants. This includes but is not limited to any pathology that would limit the blood supply to the target area or otherwise compromise healing;
6. Have a life expectancy of less than 15-months;
7. Have a history of or be planning to undergo radiotherapy in the area of the end-neuroma;
8. Have bony exostosis of the affected limb that is not treated at the time of nerve cap placement;
9. Have uncontrolled Type 1 or Type 2 Diabetes Mellitus with HbA1c of 8% or greater or those with diabetic neuropathy in the target area or proximal to the amputation site;
10. Have a history of idiopathic neuropathy/radiculopathy, known sciatica or chronic back pain;
11. Documented history of centralized nerve pain that does not respond to a peripheral nerve block in the affected limb;
12. Have a known allergy to anesthetic agents;
13. Have a known sensitivity to porcine-derived products;
14. Be currently enrolled or have been enrolled in another interventional clinical research study within the past 30 days (at time of consent); or
15. Be deemed unsuitable for inclusion in the study at the discretion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety: Adverse Events (AEs), Serious Adverse Events (SAEs), or Unanticipated Adverse Device Effects (UADEs) | 15 Months
  The primary safety endpoint will monitor the nature and incidence of AE's, SAE's and/or UADE's associated with an unplanned revision procedure prior to the planned Targeted Muscle Reinnervation (TMR) or Regenerative Peripheral Nerve Interface (RPNI) starting from implantation (operative day) through 15 months depending on whether or not the subject undergoes the secondary TMR or RPNI procedure.

SECONDARY OUTCOMES:
Change in Visual Analog Scale (VAS) For Pain Score through TMR procedure or 12 post-operative months compared to baseline | Week 2, 1, 3, 6, 9 and 12 months
  The Visual Analog Scale (VAS) For Pain is a patient reported outcomes scale whereby the patient indicates his/her current pain level by making a mark on a continuous horizontal 10-centimeter (100 millimeter) line. The distance from the 0 millimeter to the patient's mark corresponds to the amount of pain the subject is currently experiencing. VAS for Pain data are recorded as the number of millimeters from the left of the line to the patients mark across the range of 0-100 millimeters, with 0 millimeter representing no pain and 100 millimeters representing "the worst pain imaginable".
  Final VAS score will be collected either just prior to TMR or RPNI procedure or 12- months post op if subject will not undergo the secondary TMR or RPNI procedure
Change in Patient Reported Outcome Measurement Information System (PROMIS®) - Pain Related Measures through TMR or RPNI procedure or 12 post operative months compared to baseline | Week 2, 1, 3, 6, 9 and 12 months
  The Patient Reported Outcome Measurement Information System (PROMIS®) - Pain Related Measures is a set of person-centered measures that evaluates and monitors a patient's physical health and pain. The pain related measures include domains evaluating fatigue, pain intensity, pain interference, sleep Disturbance, and Pain Behavior. Short forms containing fixed sets of 4-10 items or questions are included for each domain. All PROMIS scores are presented as T-scores where the T-score is the standardized score with a mean of 50 (range 20-80) and a standard deviation of 10. Higher scores indicate more of the concept being measured where sometimes the concept is desirable (e.g., physical function) and sometimes this it is undesirable (e.g., fatigue).
  Final PROMIS® Pain Related Measure will be collected either just prior to TMR or RPNI procedure or 12-months post op if subject will not undergo the secondary TMR or RPNI procedure.
Change in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) through TMR or RPNI procedure or 12 post-operative months compared to baseline | Week 2, 1, 3, 6, 9 and 12 months
  In this study, the Work Productivity and Activity Impairment (WPAI:SHP) questionnaire is an instrument to measure impairments in both paid work and unpaid work (leisure/regular activities) due nerve injury post-surgical intervention. It measures (1) absenteeism (work time missed), (2) presenteeism (impairment at work / reduced on-the-job effectiveness), (3) work productivity loss (overall work impairment / absenteeism plus presenteeism), as well as the (4) impairments in unpaid activity because of nerve injury post-surgical intervention during the past seven days. Scores for these 4 measures are expressed as impairment percentages with higher percentage scores indicating greater impairment in than lower percentage scores.
  Final WPAI:SHP will be collected either at the office visit following the TMR or RPNI procedure or 12-months post op if subject will not undergo the secondary TMR or RPNI procedure
Change in Brief Activities Measure for Adults with Upper Limb Amputation (BAM-ULA) through 12 post-operative months compared to baseline | 3, 6, 9 and 12 months
  The BAM-ULA is a 10-item observational measure of activity performance. The 10 items are as follows: tuck a shirt in pants, lift a 20-lb bag, open a water bottle, remove a wallet from back pocket, replace the wallet in back pocket, take a gallon of water from the refrigerator and place on the counter (lift gallon jug), pour water from a gallon jug, brush or comb hair, use a fork, and open a door with knob. Items are scored with either a 0 (cannot complete all subtasks) or 1 (can complete all subtasks). Lower scores area associated with greater impairment of activity performance and higher scores are associated with less impairment of activity performance.
Change in Timed Up and Go (TUG) Test for Lower Extremity Amputees through 12 post-operative months compared to baseline | 3, 6, 9 and 12 months
  An observational test used to evaluate functional mobility in terms of postural stability, gait, stride length, and sway. Patients wear their regular footwear and can use a walking aid. They are asked to sit in a chair, stand up from that chair, walk to a line on the floor (10 ft. away) at their normal pace, turn around, walk back to the chair at a normal pace, and sit down again.
Change in the 10-Meter Walk Test (10 MWT) for Lower Extremity Amputees through 12 post-operative months compared to baseline | 3, 6, 9 and 12 months
  A performance measure used evaluate functional mobility and gait. It assesses walking speed in meters per second over 10-meter distance.
Changes in quantity and class of pain medication use at week 2, 1, 3, 6, 9, 12, and 15 post-operative months comparted to baseline | Week 2, 1, 3, 6, 9, 12, and 15 months
  Quantity and class of pain medication use for subjects who were implanted with the Axoguard Nerve Cap® will be captured during the following visits: Screening (baseline), 2-weeks, 1, 3, 6, 9, 12, and 15 months post-op for comparison to baseline.

OTHER OUTCOMES:
Nerve End Size Measurements | Prior to Secondary Surgery (if performed)
  Nerve end size as measured by MRI or CT scan prior to required secondary TMR or RPNI procedure recorded in cubic millimeters (mm3).
Histological Assessment of Explanted Nerve Cap After Secondary Procedure | Following Explant (if performed)
  Explanted tissue will be cut into thin slices, affixed to microscope slides, and stained with Hematoxylin and Eosin (H&E), Masson's Trichrome (MT) and Neurofilament 200 (NF200) to allow for histological evaluation of axonal swirling, nerve cap remodeling, and overall tissue response.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Texas Tech University, Health Science Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No